CLINICAL TRIAL: NCT02551783
Title: A Randomized Study of Dorsal Versus Ventral Buccal Mucosa Graft Onlay for Bulbar Urethroplasty
Brief Title: Dorsal vs. Ventral Buccal Graft Dorsal vs. Ventral Buccal Graft
Acronym: DoVeBuG
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Failure to recruit
Sponsor: University of Minnesota (Other)
Collaborators: University of Iowa (Other); University of Kansas (Other); Ohio State University (Other); University of Utah (Other); Loyola University Chicago (Other); Lahey Clinic (Other); University of California, San Francisco (Other); University of Washington (Other); New York University (Other); University of California, San Diego (Other); Baylor College of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1508M77183
Record Dates: First submitted 2015-08-12; First posted 2015-09-16 (Estimated); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Urethral Stricture
Keywords: urethral stricture; urethroplasty; buccal mucosa; graft
MeSH Terms: conditions — Urethral Stricture

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Urethroplasty with buccal mucosa graft (Experimental): Intervention: Procedure/Surgery: Urethroplasty with buccal graft. In this arm the graft is placed on the dorsal wall of the urethra.
  Interventions: Procedure: Urethroplasty with buccal mucosa graft
- Ventral Buccal (Active Comparator): Intervention: Procedure/Surgery: Urethroplasty with buccal graft. In this arm the graft is placed on the ventral wall of the urethra.
  Interventions: Procedure: Ventral Buccal

INTERVENTIONS:
Procedure: Urethroplasty with buccal mucosa graft — A surgery to correct urethral stricture
  Arms: Urethroplasty with buccal mucosa graft
Procedure: Ventral Buccal — Urethroplasty with buccal graft. In this arm the graft is placed on the ventral wall of the urethra.
  Arms: Ventral Buccal

SUMMARY:
This is a randomized non-blinded comparison of dorsal vs. ventral approach for buccal mucosa graft urethroplasty in the bulbar urethra. Buccal mucosa graft is a common method of repairing the strictured urethra. Current evidence suggests the two approaches for placement of the graft are equally successful at correcting the stricture and the two approaches have similar risks of complications. The investigators propose to randomly assign appropriately selected patients to either a dorsally- or ventrally-placed graft. No additional procedures beyond the normal care protocol will be required of the patients. Success will be assessed via objective and subjective methods; complications will be tallied in a standardized fashion. Outcomes will be measured at two years.

DETAILED DESCRIPTION:
Urethral strictures affect 1% of men and are rare in women. Most urethral strictures in the United States develop in the bulbar section of the urethra which is the section of the urethra proximal to the penis but distal to the prostate. A common method of surgical correction is to longitudinally open the strictured urethra and augment its width by the addition of a graft of buccal mucosa taken from the oral cavity. The urethrotomy for placement of the graft can be made along the superficial (ventral) or deep (dorsal) side of the urethra. The graft bed dorsally is the tunica albuginea of the corporal bodies (the capsule around the erectile bodies of the penis) whereas ventrally it is the corpus spongiosum of the urethra (the vascular layer that surrounds the urethra).

Ventral buccal graft onlay first described by Morey and McAninch in 1996, involves a midline perineal incision and retraction of the bulbo-spongiosum muscle downward to expose the ventral urethral surface. The corpus spongiosum is incised longitudinally to expose the urethral lumen and the incision is extended proximal and distal to the established stricture. The buccal mucosa graft is harvested and trimmed to the length and width of the urethrotomy and the graft is sutured at the proximal and distal apices and a running suture at the lateral margins to establish a tight anastomosis. Ventral placement allows for limited urethral mobilization and easy access but there is concern about higher likelihood of diverticulum formation and development of associated complications such as post-void dribbling and ejaculatory dysfunction. In addition, many surgeons have concern about graft contraction as spread-fixating the graft is not possible.

Dorsal buccal graft onlay, first described by Barbagli in 1996, also involves a midline perineal incision. The bulbo-cavernosum and corpora cavernosum are dissected from the bulbar urethra allowing for complete mobilization of the urethra. The urethra is rotated 180 degrees to allow for dorsal access and an incision is made on the dorsal urethra proximal and distal to the stricture location. The buccal graft is harvested and trimmed to the appropriate size of the urethrotomy and spread on the overlying tunica albuginea of the corporal bodies. The right mucosal margin of the urethra is sutured to the right margin of the buccal graft and the corporal bodies. The urethra is rotated back to allow for suturing of the left mucosal margin to the left margin of the buccal graft and corporal bodies, essentially covering the entire urethral plate. Dorsal placement potentially allows for a more stable vascular bed for graft sustainability and less spongiosal bleeding, but requires a greater urethral mobilization and longer operative times. The technical challenge of graft placement in a dorsal location is much greater than placement ventrally. Potential problems with dorsal placement include damage to the male external urinary sphincter, which is dorsally located, and anastomotic leakage and perineal abscess in the immediate post-operative period.

There are multiple studies that attempt to compare the outcomes of ventral versus dorsal graft placement for bulbar urethroplasty, but these studies rely on case series and retrospective data. Andrich and Mundy reported better outcomes with dorsal buccal placement, but statistical significance was not formally established. Both Barbagli and Figler were unable to demonstrate superiority of either ventral or dorsal buccal graft placement. Currently there is no high level of definitive randomized evidence to suggest superiority of either ventral or dorsal buccal placement in terms of patient outcomes and complications. In fact, the best level of evidence is VI (small case series) and dorsal vs. ventral placement is largely dependent on individual clinical judgment and comfort level with each procedure.

One factor contributing to the inability to detect a difference between dorsal vs. ventral graft placement has been the liberal definition of success that leads to uniformly high success rates across studies (85-95%) and, hence, studies that are underpowered to detect a difference in success rates. In these studies, the definition of success has typically been "need for repeat surgery". Such a definition suffers from significant detection bias in that (1) subclinical stricture recurrences may go undetected if they are not screened for; and (2) surgeon or patient reluctance to undergo a repeat surgery may lead to false negatives. When patients are rigorously followed with endoscopic inspection of the area of surgery with cystoscopy, narrowing is often identified at a much higher rate than "need for repeat surgery". For instance, in a preliminary review of our retrospective data using surveillance cystoscopy, the investigators detected narrowing in 46% of ventral buccal patients and approximately 18% of dorsal buccal patients. This more strict definition of success and the lower success rates that follow may allow for detection of a clinically meaningful difference in the success rate with the two procedures in a reasonably-sized clinical trial.

The investigators plan a randomized comparison of dorsally-placed vs. ventrally-placed buccal mucosa graft in men undergoing buccal graft urethroplasty for bulbar urethra stricture. A collaborative multi-institutional study deriving data from the Trauma and Urologic Reconstruction Network of Surgeons, a network of twelve reconstructive urology centers in the United States, would allow the investigators to achieve the required sample size within 2-3 years. The results of this study will ultimately advance research efforts in urethral stricture management and provide substantial evidence for utilization of ventral versus dorsal buccal placement for reconstructive urologists.

ELIGIBILITY:
Inclusion Criteria:

* Strictures must predominantly include the proximal and/or mid bulbar urethra and be otherwise amenable to buccal graft onlay urethroplasty
* Strictures may extend from the mid-bulbar urethra up to the distal bulbar urethra within the scrotum, but not through the scrotum to the pendulous junction
* Subjects able to consent for themselves

Exclusion Criteria:

* prior open urethral surgery, such as prior urethroplasty, artificial urinary sphincter placement, male urethral sling placement, and rectourethral fistula
* radiation therapy to the pelvis
* previous hypospadias repair
* lichen sclerosis unable to consent for themselves

Ages: 18 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Cumulative Incidence of anatomic recurrence determined by cystoscopy | 1 year
  Anatomic evidence of recurrence based on surveillance cystoscopy (i.e., if the 16F flexible cystoscope cannot bypass the surgical site then there is a failure). Flexible cystoscopy will be performed at 3 and 12 months after surgery. All surgeons will use a standard-sized scope. This will be a bivariate outcome (scope is able to pass without trauma vs. unable to pass or only able to pass with trauma)

SECONDARY OUTCOMES:
Cumulative Incidence of Complications deep venous incision and drainage | 2 years
  A composite outcome of the following rare peri-operative complications: deep venous thrombosis, positioning complaints (numbness in the feet), perineal abscess (requiring incision and drainage) and leakage of dye from the urethra on post-op voiding cystourethrogram. Each of these complications is expected to occur in about 1% of subjects. Therefore no standardized assessment will be performed: we will not perform screening ultrasound for DVT, nor will we give every patient a standardized questionnaire to assess for foot numbness. Rather, at each clinical visit, the physician will note whether the findings are present or absent based on physical exam, subjective complaints or objective tests.

OTHER OUTCOMES:
Cumulative Incidence of Secondary Procedures to Treat Stricture Recurrence restenosis | 2 years
  Occurrence of any urethral intervention for restenosis including including urethral dilation, internal urethrotomy, repeat urethroplasty, or suprapubic catheter placement.
Urinary Symptoms | 2 years
  A Patient Reported Outcome Measure (PROM) that has been validated for assessment of urinary symptoms characteristic or urethral stricture disease will be completed by patients pre-operatively and at 3, 12 and 24 months post-operatively. This asks questions about urinary hesitancy, straining, interrupted urinary stream, incomplete emptying, and post-void dribbling. Score range from 0-20 plus 2 qualitative answers. We will compare pre- and post-op as well as between dorsal and ventral graft.
Symptoms, Other pain in the penis and leakage of urine. | 2 years
  A Patient Reported Outcome Measure (PROM) that has been validated for assessment of adverse effects after urethroplasty or due to stricture itself including pain in the bladder, pain in the penis and leakage of urine. Each outcome is scored 0-3 and the outcomes are not summed. Will be completed by patients pre-operatively and at 3, 12 and 24 months post-operatively. We will compare pre- and post-op as well as between dorsal and ventral graft.
Health Status overall functioning and self-cares | 2 years
  A Patient Reported Outcome Measure (PROM) that has been validated for assessment of overall functioning and self-cares. Contains 5 questions about mobility, self-care, usual activities, pain, and anxiety/depression. There is no scoring system. Answers are not summed but are reported individually. Will be completed by patients pre-operatively and at 3, 12 and 24 months post-operatively. Will be completed by patients pre-operatively and at 3, 12 and 24 months post-operatively. We will compare pre- and post-op as well as between dorsal and ventral graft.
Evaluation of Urinary Flow | 2 years
  A Patient Reported Outcome Measure (PROM) that has been validated for assessment of urinary strength of stream in men with urethral stricture disease. This consists of a picture of the steam coming from a silhouette of a man with numbers 1-4 assigned to the stream based on how far the stream travels. Will be completed by patients pre-operatively and at 3, 12 and 24 months post-operatively. We will compare pre- and post-op as well as between dorsal and ventral graft.
Overall Health Likert scale scoring from 0-100 | 2 years
  A Likert scale scoring from 0-100 for overall health. Will be completed by patients pre-operatively and at 3, 12 and 24 months post-operatively. We will compare pre- and post-op as well as between dorsal and ventral graft.
Male Sexual Health Questionnaire | 2 years
  A PROM validated for the assessment of ejaculatory dysfunction. Has been studied some in urethroplasty patients. 4 questions with scores 0-5 are summed for a total score of 0-20. Will be completed by patients pre-operatively and at 3, 12 and 24 months post-operatively. We will compare pre- and post-op as well as between dorsal and ventral graft.
Sexual Health Inventory for Men erectile dysfunction | 2 years
  A PROM validated for the assessment of erectile dysfunction. Has been studied some in urethroplasty patients. 5 questions with scores 1-5 are summed for a total score of 5-25. Will be completed by patients pre-operatively and at 3, 12 and 24 months post-operatively. We will compare pre- and post-op as well as between dorsal and ventral graft.
Urinary Flow Rate | 2 years
  Patient urinates into a receptacle that measures the speed of his urination. Reported as maximum and mean flow rate. Will be completed by patients pre-operatively and at 3, 12 and 24 months post-operatively. We will compare pre- and post-op as well as between dorsal and ventral graft.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota Medical Center, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No